CLINICAL TRIAL: NCT02898597
Title: Smoking Cessation Intervention for Women With HIV/AIDS
Brief Title: Smoking Cessation Intervention for Women Living With HIV
Acronym: SoCIWHIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Sun S Kim, Associate Professor, University of Massachusetts, Boston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016059
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: AIDS/HIV
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video (Experimental): Video-call delivered cognitive behavioral therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Voice (Active Comparator): Voice-call delivered cognitive behavioral therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Received 8 weekly individualized counseling sessions of cognitive behavioral therapy

SUMMARY:
As people with HIV/AIDS live longer, the burden of non-AIDS-related health problems such as cardiovascular diseases and cancers on these people have consistently increased. Smoking is one of the major contributing factors to these health problems and rates of cigarette smoking in this group are substantially higher than those of the general population: 40-70% vs. 17-10%. Especially, women living with HIV/AIDS seem to be more susceptible to the negative consequence of smoking than their male counterparts. They are also less likely to see tobacco dependence treatment for dual stigma associated with both conditions: HIV infection and nicotine addiction. This is a pilot study to develop smoking cessation intervention for these women.

DETAILED DESCRIPTION:
Women are at high risk of becoming HIV positive due to biological vulnerabilities, low socioeconomic status, dominant sexual practices of males and epidemiological factors. For example, the risk of being infected with HIV during unprotected sex is two to four times greater for women than for men. With the use of combined antiretroviral therapies, these women now live longer than ever before which now faces the healthcare community with the need for evolving understanding of HIV and aging. However, the burden of non-AIDS related health problems such as cardiovascular diseases and cancers on people living with HIV/AIDS while aging has considerably increased. Smoking is one of the major contributing factors to these health problems. Rates of current cigarette smoking are substantially higher among people living with HIV/AIDS than the general population: 40-75% versus 19%. Women smokers living with HIV have a 36% higher risk for developing AIDS and 53% higher mortality when compared to non-smoking women with HIV. This study is a pilot randomized controlled trial (RCT) testing the feasibility and acceptability of a videoconferencing smoking cessation intervention (video arm) for women with HIV in comparison with a telephone-based smoking cessation intervention (telephone arm). Both arms will receive 8, 30-minute weekly cessation counseling sessions plus 8-week nicotine replacement therapy. Participants will be followed up at 1, 3 and 6 months from the target quit day. Self-reported abstinence will be verified with a saliva cotinine test using an Nicotine Alert test strip and the testing process will be monitored via mobile-phone video call.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Diagnosis of HIV infection
* Age 18 or older
* Smoking at least 5 cigarettes a day
* Having access to a mobile-phone with Internet connection
* Willing to quit smoking within the next 4 weeks

Exclusion Criteria:

* Inability to speak English
* Involvement in another cessation program
* Being pregnant or lactating
* Having an active skin disease
* History of serious mental illnesses (e.g., schizophrenia and bipolar disorder)
* Serious alcohol use problem
* Use of any illegal substances excluding marijuana

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun S Kim, PhD, Principal Investigator — University of Massachusetts, Boston
Locations (1):
- University Massachusetts Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paudel V, Baral KP. Women living with HIV/AIDS (WLHA), battling stigma, discrimination and denial and the role of support groups as a coping strategy: a review of literature. Reprod Health. 2015 Jun 2;12:53. doi: 10.1186/s12978-015-0032-9. PMID 26032304
- [Background] Bancroft A. Women, Families & HIV/AIDS: A Sociological Perspective on the Epidemic in America. J Health Psychol. 2001 May;6(3):356-8. doi: 10.1177/135910530100600309. No abstract available. PMID 22049380
- [Background] Palella FJ Jr, Baker RK, Moorman AC, Chmiel JS, Wood KC, Brooks JT, Holmberg SD; HIV Outpatient Study Investigators. Mortality in the highly active antiretroviral therapy era: changing causes of death and disease in the HIV outpatient study. J Acquir Immune Defic Syndr. 2006 Sep;43(1):27-34. doi: 10.1097/01.qai.0000233310.90484.16. PMID 16878047
- [Background] Lifson AR, Neuhaus J, Arribas JR, van den Berg-Wolf M, Labriola AM, Read TR; INSIGHT SMART Study Group. Smoking-related health risks among persons with HIV in the Strategies for Management of Antiretroviral Therapy clinical trial. Am J Public Health. 2010 Oct;100(10):1896-903. doi: 10.2105/AJPH.2009.188664. Epub 2010 Aug 19. PMID 20724677
- [Background] Minkoff H, Feldman JG, Strickler HD, Watts DH, Bacon MC, Levine A, Palefsky JM, Burk R, Cohen MH, Anastos K. Relationship between smoking and human papillomavirus infections in HIV-infected and -uninfected women. J Infect Dis. 2004 May 15;189(10):1821-8. doi: 10.1086/383479. Epub 2004 Apr 27. PMID 15122518
- [Background] Moscou-Jackson G, Commodore-Mensah Y, Farley J, DiGiacomo M. Smoking-cessation interventions in people living with HIV infection: a systematic review. J Assoc Nurses AIDS Care. 2014 Jan-Feb;25(1):32-45. doi: 10.1016/j.jana.2013.04.005. Epub 2013 Jul 20. PMID 23876816
- [Background] Vidrine DJ, Marks RM, Arduino RC, Gritz ER. Efficacy of cell phone-delivered smoking cessation counseling for persons living with HIV/AIDS: 3-month outcomes. Nicotine Tob Res. 2012 Jan;14(1):106-10. doi: 10.1093/ntr/ntr121. Epub 2011 Jun 13. PMID 21669958
- [Derived] Mdege ND, Shah S, Dogar O, Pool ER, Weatherburn P, Siddiqi K, Zyambo C, Livingstone-Banks J. Interventions for tobacco use cessation in people living with HIV. Cochrane Database Syst Rev. 2024 Aug 5;8(8):CD011120. doi: 10.1002/14651858.CD011120.pub3. PMID 39101506
- [Derived] Kim SS, DeMarco RF. The Intersectionality of HIV-Related Stigma and Tobacco Smoking Stigma With Depressive and Anxiety Symptoms Among Women Living With HIV in the United States: A Cross-sectional Study. J Assoc Nurses AIDS Care. 2022 Sep-Oct 01;33(5):523-533. doi: 10.1097/JNC.0000000000000323. Epub 2022 Jan 7. PMID 34999667
- [Derived] Kim SS, Cooley ME, Lee SA, DeMarco RF. Prediction of Smoking Abstinence in Women Living With Human Immunodeficiency Virus Infection. Nurs Res. 2020 May/Jun;69(3):167-175. doi: 10.1097/NNR.0000000000000421. PMID 31977840
- [Derived] Kim SS, Darwish S, Lee SA, Sprague C, DeMarco RF. A randomized controlled pilot trial of a smoking cessation intervention for US women living with HIV: telephone-based video call vs voice call. Int J Womens Health. 2018 Sep 25;10:545-555. doi: 10.2147/IJWH.S172669. eCollection 2018. PMID 30288127

RESULTS

PARTICIPANT FLOW:
Groups:
- Video; Telephone: Cognitive behavioral therapy Nicotine replacement therapy (Habitrol Patch)
  Cognitive Behavioral Therapy: Receive cognitive behavioral cessation counseling
Period: Overall Study
Arm/Group | Video | Telephone
Started | 25 | 24
Completed | 21 | 12
Not Completed | 4 | 12
Not completed — Protocol Violation | 4 | 2
Not completed — Lost to Follow-up | 0 | 9
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: The women who are living with HIV.
Groups:
- Video: This is the group that received the cognitive behavioral therapy for smoking cessation via video calls.
- Voice: This is the group that received the cognitive behavioral therapy for smoking cessation via voice calls.
- Total: Total of all reporting groups
Arm/Group | Video | Voice | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 22 | 47
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.76 (9.05) | 53.25 (6.49) | 50.96 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 18 | 35
  White | 2 | 1 | 3
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49
Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — The measure is based on its total score that ranges from 0 to 10. Lower scores indicate less nicotine dependence.
  units on a scale | 5.88 (2.21) | 5.16 (1.86) | 5.51 (2.05)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abstinence
Description: Self-reported abstinence since the quit day, which will be verified with a salivary cotinine test at both 3-month and 6-month follow-ups
Time Frame: 6-month follow-up
Population: Women living with HIV
Measure: Count of Participants; unit: Participants
Arm/Group | Video | Telephone
Number analyzed (Participants) | 21 | 21
Participants | 8 | 1
Statistical Analysis 1: Comparison: Video vs Telephone; Test type: Superiority; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 12.31, 95% CI 2-sided [1.37 to 110.30]
Statistical Analysis 2: Comparison: Video vs Telephone; Fisher Exact test was performed, comparing the proportion of participants whose abstinence was verified with salivary cotinine test between the two arms, which was significant (p = 0.02); Test type: Superiority; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Video | Telephone
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Video (N=25) | Telephone (N=24)
Kidney failure (Renal and urinary disorders) | 0 (0) | 1 (1) — The patient had a stroke and then diseased from kidney failure. The adverse event was not study-related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Informed Consent Form (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/97/NCT02898597/ICF_000.pdf
  • Study Protocol (2018-03-31): https://cdn.clinicaltrials.gov/large-docs/97/NCT02898597/Prot_001.pdf
  • Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/97/NCT02898597/SAP_002.pdf